CLINICAL TRIAL: NCT02416700
Title: Evaluation of Peri Implant Bone Loss of Immediately Loaded Versus Conventionally Loaded Implants With a Single Prosthesis: A Randomized and Clinical Study Split-mouth Experimental Design
Brief Title: Evaluation of Peri Implant Bone Loss of Immediately Versus Conventionally Loaded Implants With a Single Prosthesis
Acronym: Mpigozzo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mônica Nogueira Pigozzo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Mônica Nogueira Pigozzo, Student, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Mpigozzo
Record Dates: First submitted 2015-03-26; First posted 2015-04-15 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Periodontal Bone Loss
Keywords: Dental prosthesis; Patients; Osseointegrated implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate implant surgery (Experimental): Immediate implant surgery in one site.
  Interventions: Procedure: immediate implant surgery
- conventional implant surgery (Active Comparator): Conventional implant surgery in another site
  Interventions: Device: implant surgery (Straumann®)

INTERVENTIONS:
Procedure: immediate implant surgery — Surgery of dental implants in one side of the mouth.
  Other Names: surgery of dental implants
  Arms: immediate implant surgery
Device: implant surgery (Straumann®) — Dental implant surgery in one of the sides of the mouth
  Other Names: Dental implant surgery
  Arms: conventional implant surgery

SUMMARY:
The main objective of this prospective, controlled, and randomized clinical study is to evaluate the peri-implant bone loss of immediately loaded versus conventionally loaded implants with a single prosthesis. A split-mouth experimental design will be used, and the success rate of the installed implants will be determined. Twelve selected patients (corresponding to a minimum of 24 surgical implant sites) will receive endosseous Ti dental implants. The protocol for preparing the surgical sites will be based on the manufacturer's recommendations and bone density. Patients with an initial torque less than 30 N·cm and an implant stability quotient (ISQ) less than 60 will be excluded from the research. Envelopes, indicating which site is the test site, will be opened after the implants are installed. Transfer impressions of the implants receiving immediate loading will be produced so that temporary crowns can be made. Temporary crowns will be installed a maximum of 24 hours after the surgery, by using the torque recommended by the manufacturer. Appropriate occlusal adjustment will be made to ensure minimal contact at maximum intercuspation and absence of contacts during protrusive and lateral excursive movements of the jaw. At baseline (time of implant installation) and 3, 6, 9, and 12 months after implant installation, the following aspects will be evaluated: the initial torque at the moment of implant insertion, Osstell ISQ, pain in the implant when subjected to vertical and horizontal forces, clinical mobility of the implant, crestal bone loss around the implant (as determined by x-ray evaluation), probing depth around the implant, and periodontal pain.

DETAILED DESCRIPTION:
The main objective of this prospective, controlled, and randomized clinical study is to evaluate the peri-implant bone loss of immediately loaded versus conventionally loaded implants with a single prosthesis. A split-mouth experimental design will be used, and the success rate of the installed implants will be determined. Twelve selected patients (corresponding to a minimum of 24 surgical implant sites) will receive endosseous Ti dental implants. The protocol for preparing the surgical sites will be based on the manufacturer's recommendations and bone density. Patients with an initial torque less than 30 N·cm and an implant stability quotient (ISQ) less than 60 will be excluded from the research. Envelopes, indicating which site is the test site, will be opened after the implants are installed. Transfer impressions of the implants receiving immediate loading will be produced so that temporary crowns can be made. Temporary crowns will be installed a maximum of 24 hours after the surgery, by using the torque recommended by the manufacturer. Appropriate occlusal adjustment will be made to ensure minimal contact at maximum intercuspation and absence of contacts during protrusive and lateral excursive movements of the jaw. At baseline (time of implant installation) and 3, 6, 9, and 12 months after implant installation, the following aspects will be evaluated: the initial torque at the moment of implant insertion, Osstell ISQ, pain in the implant when subjected to vertical and horizontal forces, clinical mobility of the implant, crestal bone loss around the implant (as determined by x-ray evaluation), probing depth around the implant, and periodontal pain. These data will be collected for both the control/delayed loading group and the test/immediate loading group, followed by statistical analysis

ELIGIBILITY:
Inclusion Criteria: edentulous sites bilateral in maxilla and mandibula with adequate quantity of bone

Exclusion Criteria: Patients with an initial torque less than 30 N·cm and an implant stability quotient (ISQ) less than 60 will be excluded from the research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Bone Loss of Immediate Versus Conventional Implants as determined by x-ray evaluation | 12 months
  The same bone loss of for conventional and immediate implants.

SECONDARY OUTCOMES:
The success rate of the installed implants will be determined | 12 months
  Survival rate must be the same for the immediate and conventional implants

CONTACTS AND LOCATIONS:
Overall Officials: Mônica N. Pigozzo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Mônica Nogueira Pigozzo, São Paulo, Brazil

REFERENCES:
- [Background] Galindo-Moreno P, Leon-Cano A, Ortega-Oller I, Monje A, O Valle F, Catena A. Marginal bone loss as success criterion in implant dentistry: beyond 2 mm. Clin Oral Implants Res. 2015 Apr;26(4):e28-e34. doi: 10.1111/clr.12324. Epub 2014 Jan 3. PMID 24383987
- [Background] Cannizzaro G, Felice P, Leone M, Ferri V, Viola P, Esposito M. Immediate versus early loading of 6.5 mm-long flapless-placed single implants: a 4-year after loading report of a split-mouth randomised controlled trial. Eur J Oral Implantol. 2012 Summer;5(2):111-21. PMID 22866288
- See also: Galindo-Moreno P, León-Cano A, Ortega-Oller I, Monje A, O Valle F, Catena A. Marginal bone loss as success criterion in implant dentistry: beyond 2 mm. — http://www.ncbi.nlm.nih.gov/pubmed/24383987